CLINICAL TRIAL: NCT04323969
Title: Foot Progression Angle Modification: an Exploratory Six-week Intervention in People With Knee Osteoarthritis
Brief Title: Gait Modification for Knee Osteoarthritis
Acronym: SENSMOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-related laboratory shutdown.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Hunt, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H19-02621
Record Dates: First submitted 2020-02-03; First posted 2020-03-27 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Gait Modification; Wearable Sensors
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Modification Target (Experimental): A 15 degree relative increase to foot progression angle
  Interventions: Behavioral: Specific Modification Target
- Self-directed Modification (Experimental): A self-directed increase to foot progression angle that is "as much as is comfortable".
  Interventions: Behavioral: Self-directed Modification

INTERVENTIONS:
Behavioral: Specific Modification Target — Participants will be instructed to increase their baseline foot progression angle by 15 degrees. Visual feedback during practice will be delivered using a mirror and guideline (tape placed on mirror). Verbal feedback will be incorporated to encourage participants to perform the modified foot progression angle as accurately as possible.
  Arms: Specific Modification Target
Behavioral: Self-directed Modification — Participants will be instructed to modify their foot progression angle as much as is comfortable. A mirror will be used during practice for visual feedback, but no specific target or guide will be provided.
  Arms: Self-directed Modification

SUMMARY:
This randomized clinical trial will compare the changes in performance, biomechanical and clinical outcomes before and after a six-week gait modification intervention. Participants with knee osteoarthritis will attend in-lab assessments and practice, while also performing daily, at-home walking tracked using a custom sensorized shoe.

DETAILED DESCRIPTION:
Greater toe-in or toe-out angles during walking are potential biomechanical management strategies for medial compartment knee osteoarthritis (OA). Multi-week clinical trials demonstrate the biomechanical efficacy and potential clinical efficacy. However, walking biomechanics have only been assessed within laboratory environments and performance of the modifications during daily at-home walking is currently unknown. Furthermore, the modifications have largely been instructed using a specific target, requiring motor learning. No study has examined whether a self-directed strategy is feasible and will produce significant improvements in biomechanical and clinical outcomes. Moreover, objective real-world performance of these modifications is unknown and may explain the previous inconsistent clinical results. This study will address these gaps. The investigators hypothesize that real-world performance of the modifications will improve over the intervention and that both groups will exhibit improvements in biomechanical and clinical outcomes at follow up.

ELIGIBILITY:
Inclusion Criteria:

* Be 50 years of age or greater
* Exhibit signs of tibiofemoral OA (a score of ≥ 2 on the Kellgren and Lawrence (KL) grading scale) predominantly in the medial compartment,
* Self-reported knee pain ≥ 3 / 10 on a numerical rating scale of pain (NRS; 0 = "no pain" and 10 = "worst pain imaginable") during most days of the previous month
* Are comfortable walking intermittently for 30 minutes
* Fit into the available sizes of sensorized shoes (sizes spanning US women's 5 to men's 13)
* Exhibit at least a 5% reduction in knee adduction moment impulse for 10 degrees of change to foot rotation measured during a screening appointment.

Exclusion Criteria:

* Any knee surgery or intraarticular injections within the past 6 months
* A history of joint replacement surgery or high tibial osteotomy
* Current or recent (within 6 weeks) corticosteroid injections
* Use of a gait aid
* Currently on a wait list for joint replacement surgery or high tibial osteotomy
* Any inflammatory arthritic condition
* Any other conditions that may affect normal gait or participation in an aerobic exercise program
* Cannot attend all required appointments.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Change in baseline to week 7 foot rotation angle error during stance - in lab walking | Baseline, Week 7
  Foot rotation is the specific walking parameter that will be modified during the intervention. It is defined as the angle between the long axis of the foot (heel to toe) and the walking direction. Foot rotation will be measured via standard marker-based motion capture and sensor-based motion capture during baseline, follow up, and each practice session.
Weekly change in baseline foot rotation angle error during stance - at home walking and during practice sessions | Baseline, Weeks 1, 2, 3, 4, 5, 6, 7
  Foot rotation is the specific walking parameter that will be modified during the intervention. It is defined as the angle between the long axis of the foot and the walking direction. Foot rotation will be measured via sensor-based motion capture over each week of the intervention. Median and inter-quartile ranges will be taken as the primary summary statistic.

SECONDARY OUTCOMES:
Change in baseline to week 7 knee joint moment impulse | Baseline, Week 7
  Knee flexion and adduction moment impulses will be calculated. Participants will walk on an instrumented walkway (2 force platforms) while 14 high speed cameras track the trajectories of markers placed on boney landmarks. Moments will be calculated using an inverse dynamics approach.
Change in baseline to week 7 Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, Week 7
  Validated questionnaire on symptoms and functional limitations related to knee osteoarthritis. The score is expressed in percentage (0-100), with 0 representing extreme knee problems and 100 representing no knee problems.
Change in baseline to week 7 knee pain on a numerical rating scale | Baseline, Week 7
  Knee pain rated on a 0 to 10 scale. 0 = "no pain at all" and 10 = "worst pain imaginable".
Change in week 1 to week 7 difficulty performing the modification on a numerical rating scale | Week 1, 7
  Difficulty will be rated on a 0 to 10 scale. 0 = "no difficulty at all" and 10 = "most difficulty imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hunt, PT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Motion Analysis and Biofeedback Laboratory, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04323969/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04323969/SAP_001.pdf